CLINICAL TRIAL: NCT01715285
Title: A Randomized, Double-blind, Comparative Study of Abiraterone Acetate Plus Low-Dose Prednisone Plus Androgen Deprivation Therapy (ADT) Versus ADT Alone in Newly Diagnosed Subjects With High-Risk, Metastatic Hormone-naive Prostate Cancer (mHNPC)
Brief Title: A Study of Abiraterone Acetate Plus Low-Dose Prednisone Plus Androgen Deprivation Therapy (ADT) Versus ADT Alone in Newly Diagnosed Participants With High-Risk, Metastatic Hormone-Naive Prostate Cancer (mHNPC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100900; 212082PCR3011 (Other: Janssen Research & Development, LLC); 2012-002940-26 (EudraCT Number); U1111-1135-7146 (Other: Universal Trial Number)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Prostate cancer; Metastatic prostate cancer; Abiraterone acetate; ZYTIGA; Prednisone; Androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Abiraterone acetate + Prednisone + ADT (Experimental): Participants will receive abiraterone acetate tablet at a total dose of 1000 milligram (mg) plus 5 mg capsule of prednisone orally once daily until disease progression, withdrawal of consent or unacceptable toxicity. Stable regimen of androgen deprivation therapy (ADT) will be administered.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Other: Androgen deprivation therapy (ADT)
- Placebo + Androgen Deprivation Therapy (ADT) (Placebo Comparator): Participants will receive placebo matched to abiraterone acetate plus prednisone orally once daily until disease progression, withdrawal of consent or unacceptable toxicity. Stable regimen of ADT will be administered.
  Interventions: Other: Androgen deprivation therapy (ADT); Drug: Abiraterone acetate Placebo; Drug: Prednisone Placebo

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate tablets will be administered orally at a total dose of 1000 mg per day until disease progression, withdrawal of consent or unacceptable toxicity.
  Other Names: Zytiga
  Arms: Abiraterone acetate + Prednisone + ADT
Drug: Prednisone — Prednisone 5 mg capsule will be administered orally once daily until disease progression, withdrawal of consent or unacceptable toxicity.
  Arms: Abiraterone acetate + Prednisone + ADT
Other: Androgen deprivation therapy (ADT) — All participants will receive stable regimen of ADT, that is, lutenizing hormone releasing hormone (LHRH) agonists or surgical castration according to local guidelines until disease progression, withdrawal of consent or unacceptable toxicity.
Drug: Abiraterone acetate Placebo — Placebo matched to abiraterone acetate will be administered orally once daily until disease progression, withdrawal of consent or unacceptable toxicity.
  Arms: Placebo + Androgen Deprivation Therapy (ADT)
Drug: Prednisone Placebo — Placebo matched to prednisone will be administered orally once daily until disease progression, withdrawal of consent or unacceptable toxicity.
  Arms: Placebo + Androgen Deprivation Therapy (ADT)

SUMMARY:
The purpose of this study is to determine if newly diagnosed (within previous 3 months) participants with metastatic (spread of cancer cells from one part of the body to another ) hormone-naive prostate cancer (mHNPC) who have high-risk prognostic factors will benefit from the addition of abiraterone acetate plus low-dose prednisone to androgen deprivation therapy (ADT; lutenizing hormone releasing hormone [LHRH] agonists or surgical castration).

DETAILED DESCRIPTION:
This is a randomized (the treatment group is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study designed to determine the efficacy of abiraterone acetate plus low-dose prednisone in participants with mHNPC. The study consists of 4 parts: Screening Phase (that is, 28 days before study commences on Day 1); Double-blind treatment Phase (consists of 4-week dosing cycles wherein abiraterone acetate will be administered as 1,000 milligram [mg] plus 5 mg prednisone or only placebo orally); Follow-up Phase (every 4 months up to 60 months or until death, lost to follow up, withdrawal of consent or study termination) Open-label Extension (OLE) Phase. Participants in the Double-blind Treatment Phase will have the opportunity to enroll into the OLE Phase. The OLE Phase will allow participants to receive active drug (abiraterone acetate plus prednisone) until Long-term Extension (LTE) Phase for an additional period of up to 3 years. Participants will discontinue study treatment at disease progression or unacceptable toxicity unless, in the Investigator's opinion, it is deemed that the participants will continue to derive benefit from study treatment. Participants will be randomized in a 1:1 ratio to the active treatment group (abiraterone acetate 1000 mg daily plus prednisone 5 mg daily plus ADT) or the control group (ADT plus placebos).Efficacy will be evaluated primarily by overall survival and radiographic progression-free survival. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic prostate cancer within 3 months prior to randomization with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Distant metastatic disease documented by positive bone scan or metastatic lesions on computed tomography (CT) or magnetic resonance imaging (MRI) scan
* At least 2 of the following high-risk prognostic factors: Gleason score of greater than or equal to (>=8); presence of 3 or more lesions on bone scan; presence of measurable visceral (excluding lymph node disease) metastasis on CT or MRI Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 scan
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0, 1 or 2
* Adequate hematologic, hepatic, and renal function
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone use contraindicated
* Any chronic medical condition requiring a higher systemic dose of corticosteroid than 5 mg prednisone per day
* Pathological finding consistent with small cell carcinoma of the prostate
* Known brain metastasis
* Any prior pharmacotherapy, radiation therapy, or surgery for metastatic prostate cancer (the following exception are permitted): up to 3 months of androgen deprivation therapy (ADT) with lutenizing hormone releasing hormone agonists or antagonists or orchiectomy with or without concurrent anti-androgens prior Cycle 1 Day 1; participants may have one course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease if it was administered at least 28 days prior to Cycle 1 Day 1)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1209 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2022-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (208):
- Argentina (5):
  - Buenos Aires
  - Caba
  - Córdoba
  - La Rioja
  - Rosario
- Australia (6):
  - Adelaide
  - Footscray
  - Liverpool
  - Malvern
  - Randwick
  - Wahroonga
- Belgium (10):
  - Antwerp
  - Bonheiden
  - Brasschaat
  - Brussels
  - Charleroi
  - Liège
  - Namur
  - Ottignies
  - Sint-Niklaas
  - Yvoir
- Brazil (14):
  - Barretos
  - Belo Horizonte
  - Caxias do Sul
  - Curitiba
  - Ijuí
  - Jaú
  - Natal
  - Novo Hamburgo
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - São José do Rio Preto
  - São Paulo
- Bulgaria (2):
  - Gabrovo
  - Sofia
- Canada (10):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Kingston, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Santiago, Chile
- China (10):
  - Beijing
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Suzhou
  - Tianjin
  - Wuhan
- Colombia (3):
  - Bogotá
  - Floridablanca
  - Medellín
- Czechia (4):
  - Hradec Králové
  - Olomouc
  - Pilsen
  - Prague
- Denmark (5):
  - Aarhus N
  - Holsterbro
  - Odense
  - Roskilde
  - Vejle
- Finland (2):
  - Oulu
  - Tampere
- France (7):
  - La Chaussée-Saint-Victor
  - Lille
  - Montpellier
  - Paris
  - Suresnes
  - Toulouse
  - Villejuif
- Germany (3):
  - Düsseldorf
  - Hamburg
  - Nürtingen
- Hungary (5):
  - Budapest
  - Győr
  - Miskolc
  - Pécs
  - Szentes
- Israel (7):
  - Beer Yaakov
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
- Japan (12):
  - Chiba
  - Gifu
  - Kashiwa
  - Matsuyama
  - Nankoku
  - Ōsaka-sayama
  - Sakura
  - Tokushima
  - Tokyo
  - Ube
  - Yokohama
  - Yufu
- Malaysia (2):
  - Kuala Lumpur
  - Kuching
- Mexico (8):
  - Chihuahua City
  - Cuernavaca
  - Durango
  - Guadalajara
  - Monterrey
  - Oaxaca City
  - Pachuca
  - Zapopan
- Netherlands (7):
  - Alkmaar
  - Amsterdam
  - Amsterdam-Zuidoost
  - Hilversum
  - Hoofddorp
  - Nieuwegein
  - Rotterdam
- New Zealand (4):
  - Auckland
  - Christchurch
  - Hamilton
  - Tauranga
- Poland (5):
  - Bydgoszcz
  - Gdansk
  - Lodz
  - Lublin
  - Warsaw
- Portugal (4):
  - Braga
  - Coimbra
  - Lisbon
  - Porto
- Romania (4):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Iași
- Russia (21):
  - Chelyabinsk
  - Ivanovo
  - Izhevsk
  - Moscow
  - Nizhny Novgorod
  - Obninsk
  - Omsk
  - Orenburg
  - Pyatigorsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Saransk
  - Saratov
  - Sochi
  - Stavropol
  - Tyumen
  - Ufa
  - Volgograd
  - Yekaterinburg
  - Yoshkar-Ola
- Slovakia (6):
  - Košice-Šaca
  - Martin
  - Piešťany
  - Prešov
  - Rimavská Sobota
  - Trnava
- South Africa (4):
  - George
  - Port Elizabeth
  - Pretoria
  - Vosloorus
- South Korea (6):
  - Bucheon-si
  - Busan
  - Daegu
  - Daejeon
  - Gyeonggi-do
  - Seoul
- Spain (5):
  - A Coruña
  - Barcelona
  - Córdoba
  - Madrid
  - Murcia
- Sweden (5):
  - Gothenburg
  - Malmo
  - Stockholm
  - Umeå
  - Uppsala
- Turkey (Türkiye) (5):
  - Adana
  - Ankara
  - Istanbul
  - Izmir
  - Zonguldak
- Ukraine (10):
  - Cherkassy
  - Dnipro
  - Khakhiv
  - Kharkiv
  - Kyiv
  - Lviv
  - Makiivka
  - Odesa
  - Uzhhorod
  - Zaporizhzhia
- United Kingdom (6):
  - Cambridge
  - Glasgow
  - Manchester
  - Nottingham
  - Oxford
  - Plymouth

REFERENCES:
- [Derived] Koroki Y, Taguri M. Clinical Outcomes of First Subsequent Therapies After Abiraterone Acetate Plus Prednisone for High-Risk Metastatic Castration-Sensitive Prostate Cancer in the LATITUDE Study. Target Oncol. 2023 Jan;18(1):119-128. doi: 10.1007/s11523-022-00929-3. Epub 2022 Nov 28. PMID 36443540
- [Derived] Koroki Y, Taguri M, Matsubara N, Fizazi K. Estimation of Overall Survival with Subsequent Treatment Effect by Applying Inverse Probability of Censoring Weighting in the LATITUDE Study. Eur Urol Open Sci. 2022 Jan 6;36:51-58. doi: 10.1016/j.euros.2021.11.012. eCollection 2022 Feb. PMID 35098170
- [Derived] Baciarello G, Ozguroglu M, Mundle S, Leitz G, Richarz U, Hu P, Feyerabend S, Matsubara N, Chi KN, Fizazi K. Impact of abiraterone acetate plus prednisone in patients with castration-sensitive prostate cancer and visceral metastases over four years of follow-up: A post-hoc exploratory analysis of the LATITUDE study. Eur J Cancer. 2022 Feb;162:56-64. doi: 10.1016/j.ejca.2021.11.026. Epub 2021 Dec 23. PMID 34953443
- [Derived] Azad AA, Armstrong AJ, Alcaraz A, Szmulewitz RZ, Petrylak DP, Holzbeierlein J, Villers A, Alekseev B, Iguchi T, Shore ND, Gomez-Veiga F, Rosbrook B, Lee HJ, Haas GP, Stenzl A. Efficacy of enzalutamide in subgroups of men with metastatic hormone-sensitive prostate cancer based on prior therapy, disease volume, and risk. Prostate Cancer Prostatic Dis. 2022 Feb;25(2):274-282. doi: 10.1038/s41391-021-00436-y. Epub 2021 Aug 21. PMID 34420037
- [Derived] Feyerabend S, Saad F, Perualila NJ, Van Sanden S, Diels J, Ito T, De Porre P, Fizazi K. Adjusting Overall Survival Estimates for Treatment Switching in Metastatic, Castration-Sensitive Prostate Cancer: Results from the LATITUDE Study. Target Oncol. 2019 Dec;14(6):681-688. doi: 10.1007/s11523-019-00685-x. PMID 31754962
- [Derived] Fizazi K, Tran N, Fein L, Matsubara N, Rodriguez-Antolin A, Alekseev BY, Ozguroglu M, Ye D, Feyerabend S, Protheroe A, Sulur G, Luna Y, Li S, Mundle S, Chi KN. Abiraterone acetate plus prednisone in patients with newly diagnosed high-risk metastatic castration-sensitive prostate cancer (LATITUDE): final overall survival analysis of a randomised, double-blind, phase 3 trial. Lancet Oncol. 2019 May;20(5):686-700. doi: 10.1016/S1470-2045(19)30082-8. Epub 2019 Apr 12. PMID 30987939
- [Derived] Li T, Franco-Villalobos C, Proskorovsky I, Sorensen SV, Tran N, Sulur G, Chi KN. Medical resource utilization of abiraterone acetate plus prednisone added to androgen deprivation therapy in metastatic castration-naive prostate cancer: Results from LATITUDE. Cancer. 2019 Feb 15;125(4):626-632. doi: 10.1002/cncr.31847. Epub 2018 Dec 6. PMID 30521063
- [Derived] Chi KN, Protheroe A, Rodriguez-Antolin A, Facchini G, Suttman H, Matsubara N, Ye Z, Keam B, Damiao R, Li T, McQuarrie K, Jia B, De Porre P, Martin J, Todd MB, Fizazi K. Patient-reported outcomes following abiraterone acetate plus prednisone added to androgen deprivation therapy in patients with newly diagnosed metastatic castration-naive prostate cancer (LATITUDE): an international, randomised phase 3 trial. Lancet Oncol. 2018 Feb;19(2):194-206. doi: 10.1016/S1470-2045(17)30911-7. Epub 2018 Jan 8. PMID 29326030
- [Derived] Fizazi K, Tran N, Fein L, Matsubara N, Rodriguez-Antolin A, Alekseev BY, Ozguroglu M, Ye D, Feyerabend S, Protheroe A, De Porre P, Kheoh T, Park YC, Todd MB, Chi KN; LATITUDE Investigators. Abiraterone plus Prednisone in Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2017 Jul 27;377(4):352-360. doi: 10.1056/NEJMoa1704174. Epub 2017 Jun 4. PMID 28578607

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1209 participants were enrolled and 1199 were randomized to treatment groups.10 participants from Russian site were excluded from the analysis due to noncompliance with International Conference on Harmonization Good Clinical Practice guidelines at site. The remaining 1199 randomized participants comprised the intent-to-treat population.
Groups:
- Abiraterone Acetate+Prednisone+ADT: Participants received abiraterone acetate tablet at a total dose of 1000 milligram (mg) plus 5 mg capsule of prednisone orally once daily until disease progression, withdrawal of consent or unacceptable toxicity. Stable regimen of androgen deprivation therapy (ADT) was administered.
- Placebo + ADT: Participants received placebo matched to abiraterone acetate plus prednisone orally once daily until disease progression, withdrawal of consent or unacceptable toxicity. Stable regimen of ADT was administered.
- DB Period Placebo to Open-label Extension (OLE) Abiraterone Acetate: Participants who were originally randomized to the Placebo group were permitted to crossover to Abiraterone Acetate plus Prednisone treatment in open-label extension phase to receive abiraterone acetate tablet at a total dose of 1000 mg plus 5 mg capsule of prednisone orally once daily until disease progression, withdrawal of consent or unacceptable toxicity.
Period: Double Blind Period (Up to 23 Months)
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT | DB Period Placebo to Open-label Extension (OLE) Abiraterone Acetate
Started | 597 | 602 | 0
Completed | 0 | 0 | 0
Not Completed | 597 | 602 | 0
Not completed — Adverse Event | 53 | 31 | 0
Not completed — Death | 43 | 25 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Physician Decision | 21 | 23 | 0
Not completed — Withdrawal by Subject | 52 | 47 | 0
Not completed — Progressive Disease | 254 | 388 | 0
Not completed — Noncompliance With Study Drug | 4 | 2 | 0
Not completed — Placebo Cross-Over | 0 | 72 | 0
Not completed — Other | 167 | 12 | 0
Period: OLE Phase (Up to 15.6 Months)
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT | DB Period Placebo to Open-label Extension (OLE) Abiraterone Acetate
Started | 0 | 0 | 72 (Post unblinding, participants crossed over to OLE Phase.)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 72
Not completed — Death | 0 | 0 | 4
Not completed — Other | 0 | 0 | 60
Not completed — Progressive Disease | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) analysis set included all participants randomized into the study and who were classified according to their assigned treatment group, regardless of the actual treatment received. .
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT | Total
Number analyzed (Participants) | 597 | 602 | 1199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years: <=18 years | 0 | 0 | 0
  <=18 years: Between 18 and 65 years | 221 | 233 | 454
  <=18 years: >=65 years | 376 | 369 | 745
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8.48) | 66.8 (8.72) | 67.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 597 | 602 | 1199
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 8 | 8 | 16
  Australia | 4 | 4 | 8
  Belgium | 6 | 7 | 13
  Brazil | 28 | 28 | 56
  Bulgaria | 1 | 1 | 2
  Canada | 16 | 17 | 33
  Chile | 3 | 4 | 7
  China | 69 | 68 | 137
  Colombia | 10 | 7 | 17
  Czech Republic | 9 | 7 | 16
  Denmark | 13 | 15 | 28
  Finland | 4 | 5 | 9
  France | 7 | 7 | 14
  Germany | 4 | 4 | 8
  Hungary | 17 | 17 | 34
  Israel | 14 | 16 | 30
  Italy | 19 | 20 | 39
  Japan | 35 | 35 | 70
  Malaysia | 4 | 2 | 6
  Mexico | 19 | 19 | 38
  Netherlands | 6 | 4 | 10
  New Zeland | 6 | 5 | 11
  Poland | 20 | 22 | 42
  Portugal | 19 | 20 | 39
  Romania | 22 | 21 | 43
  Russian Federation | 89 | 95 | 184
  Slovakia | 17 | 14 | 31
  South Africa | 10 | 10 | 20
  South Korea | 16 | 16 | 32
  Spain | 16 | 17 | 33
  Sweden | 11 | 11 | 22
  Turkey | 18 | 17 | 35
  Ukraine | 39 | 40 | 79
  United Kingdom | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-Free Survival (PFS)
Description: Radiographic PFS was defined as the time (in months) interval from randomization to the first date of radiographic progression or death. Radiographic progression included progression by bone scan (according to modified Prostate Cancer Working Group 2 [PCWG2] criteria), defined as at least 2 new lesions on bone scan and progression of soft tissue lesions by computed tomography (CT) or magnetic resonance imaging (MRI) (according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria). As per the RECIST 1.1 guideline, progression requires a 20 percent (%) increase in the sum of diameters of all target lesions and a minimum absolute increase of 5 millimeter (mm) in the sum as compared to nadir sum of diameter.
Time Frame: Up to 44 months
Population: Intention to treat (ITT) analysis set included all subjects randomized into the study and who were classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT
Number analyzed (Participants) | 597 | 602
Months | 33.02 [29.57 to NA] — Here 'NA' represents that upper limit of 95% CI was not estimable due to lesser number of events. | 14.78 [14.69 to 18.27]
Statistical Analysis 1: Comparison: Abiraterone Acetate+Prednisone+ADT vs Placebo + ADT; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.466, 95% CI 2-sided [0.394 to 0.550]

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to date of death from any cause.
Time Frame: Up to 66 months
Population: ITT analysis set included all subjects randomized into the study and who were classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT
Number analyzed (Participants) | 597 | 602
months | 53.32 [48.23 to NA] — Here 'NA' represents that upper limit of 95% CI was not estimable due to lesser number of events. | 36.53 [33.54 to 39.95]
Statistical Analysis 1: Comparison: Abiraterone Acetate+Prednisone+ADT vs Placebo + ADT; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.661, 95% CI 2-sided [0.564 to 0.775]

3. Secondary Outcome: Time to Initiation of Chemotherapy
Description: Time to initiation of chemotherapy was defined as the time (in months) interval from the date of randomization to the date of initiation of cytotoxic chemotherapy for prostate cancer.
Time Frame: Up to 66 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT
Number analyzed (Participants) | 597 | 602
months | NA [62.62 to NA] — Here, 'NA' indicates that the median and upper limit of 95% CI was not estimated due to lesser number of events. | 57.59 [38.18 to NA] — Here, 'NA' indicates that the upper limit of 95% CI was not estimated due to lesser number of events.

4. Secondary Outcome: Time to Subsequent Therapy for Prostate Cancer
Description: Time to subsequent therapy was defined as the time (in months) interval from the date of randomization to the date of initiation of subsequent therapy for prostate cancer.
Time Frame: Up to 66 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT
Number analyzed (Participants) | 597 | 602
Months | 54.87 [46.42 to NA] — Here 'NA' indicates that the upper limit of 95% CI was not estimated due to lesser number of events. | 21.22 [18.56 to 23.49]

5. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the time (in months) interval from randomization to the first date a participant experienced a greater than or equal to (>=) 30 percent (%) increase in Brief Pain Inventory-Short Form (BPI-SF) from baseline in the BPI-SF worst pain intensity (Item 3) observed at 2 consecutive evaluations (>=4) weeks apart. BPI-SF was an 11-item questionnaire, designed to assess severity and impact of pain on daily functions. Total score ranged from 0 to 10 with 0 representing "no pain" and 10 representing" pain as bad as you can imagine.
Time Frame: Up to 66 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT
Number analyzed (Participants) | 597 | 602
Months | 47.41 [33.15 to NA] — Here 'NA' represents that upper limit of 95% CI was not estimable due to lesser number of events. | 16.62 [11.07 to 23.95]

6. Secondary Outcome: Time to Skeletal-Related Event
Description: Time to skeletal-related event was defined as the earliest of the following: clinical or pathological fracture, spinal cord compression, palliative radiation to bone, or surgery to bone.
Time Frame: Up to 66 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT
Number analyzed (Participants) | 597 | 602
months | NA [NA to NA] — Here 'NA' represents that median, upper limit and lower limit of 95% CI was not estimable due to lesser number of events. | NA [NA to NA] — Here 'NA' represents that median, upper limit and lower limit of 95% CI was not estimable due to lesser number of events.

7. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as the time (in months) interval from the date of randomization to the date of PSA progression, according to PCWG2 criteria. PCWG2 defines PSA progression as the date that a 25 percent (%) or greater increase and an absolute increase of 2 nanogram per milliliter (ng/mL) or more from the nadir is documented, which is confirmed by a second value obtained 3 or more weeks later.
Time Frame: Up to 66 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT
Number analyzed (Participants) | 597 | 602
Months | 33.31 [29.44 to 46.09] | 7.43 [7.20 to 9.20]

ADVERSE EVENTS:
Time Frame: From Day 1 up to 30 days post last dose (that is, for DB period: up to 23 months and OLE period: up to 15.6 months), deaths were collected from baseline up to end of study (up to 66 months).
Description: Safety analysis set included all participants randomized into the study and who received any part of study drug. Only 72 deaths out of all cause mortalities contributed to discontinuation.
Arm/Group | Abiraterone Acetate+Prednisone+ADT | Placebo + ADT | DB Period Placebo to Open-label Extension (OLE) Abiraterone Acetate
All-Cause Mortality (participants affected / at risk) | 275/597 | 339/602 | 4/72
Serious Adverse Events (participants affected / at risk) | 192/597 | 151/602 | 4/72
Other Adverse Events (participants affected / at risk) | 533/597 | 515/602 | 35/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate+Prednisone+ADT (N=597) | Placebo + ADT (N=602) | DB Period Placebo to Open-label Extension (OLE) Abiraterone Acetate (N=72)
Anaemia (Blood and lymphatic system disorders) | 6 | 6 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 5 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 3 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 0
Atrial Flutter (Cardiac disorders) | 2 | 0 | 0
Cardiac Failure (Cardiac disorders) | 3 | 0 | 0
Cardiac Failure Acute (Cardiac disorders) | 2 | 0 | 0
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 3 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 1 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Abdominal Mass (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal Polyp (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Device Dislocation (General disorders) | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 2 | 1 | 0
Hernia Pain (General disorders) | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 2 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 3 | 0
Peripheral Swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 6 | 2 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatobiliary Disease (Hepatobiliary disorders) | 1 | 0 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 0
Bronchopneumonia (Infections and infestations) | 3 | 1 | 0
Bursitis Infective (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cellulitis Orbital (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Eye Infection (Infections and infestations) | 1 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 2 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Localised Infection (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis Acute (Infections and infestations) | 0 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 12 | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 2 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Spinal Cord Infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 8 | 5 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Kidney Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 0 | 0
Biopsy Liver (Investigations) | 1 | 0 | 0
Blood Glucose Abnormal (Investigations) | 0 | 1 | 0
Blood Testosterone Increased (Investigations) | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Metabolic Syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 10 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic Lymphocytic Leukaemia Stage 3 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lentigo Maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Neoplasm of Renal Pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm of Thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 1 | 0
Brain Compression (Nervous system disorders) | 0 | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 2 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 3 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 1 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 1 | 0
Lacunar Infarction (Nervous system disorders) | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 2 | 0 | 0
Myasthenia Gravis (Nervous system disorders) | 0 | 1 | 0
Nerve Compression (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Optic Nerve Compression (Nervous system disorders) | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 3 | 0
Paraplegia (Nervous system disorders) | 2 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0
Speech Disorder (Nervous system disorders) | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 11 | 11 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 2 | 1 | 0
Vascular Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Mental Disorder (Psychiatric disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2 | 0
Bladder Outlet Obstruction (Renal and urinary disorders) | 0 | 1 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 2 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 2 | 0
Haematuria (Renal and urinary disorders) | 8 | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 2 | 0
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 1 | 2 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0
Renal Failure (Renal and urinary disorders) | 3 | 1 | 0
Renal Injury (Renal and urinary disorders) | 1 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urethral Haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 10 | 11 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 3 | 3 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lipoma Excision (Surgical and medical procedures) | 1 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0 | 0
Aortic Dissection (Vascular disorders) | 0 | 1 | 0
Blood Pressure Fluctuation (Vascular disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 4 | 4 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 2 | 0
Hypertensive Crisis (Vascular disorders) | 2 | 0 | 0
Intermittent Claudication (Vascular disorders) | 2 | 0 | 0
Peripheral Vascular Disorder (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate+Prednisone+ADT (N=597) | Placebo + ADT (N=602) | DB Period Placebo to Open-label Extension (OLE) Abiraterone Acetate (N=72)
Anaemia (Blood and lymphatic system disorders) | 58 | 89 | 3
Abdominal Pain (Gastrointestinal disorders) | 26 | 31 | 0
Constipation (Gastrointestinal disorders) | 68 | 67 | 2
Diarrhoea (Gastrointestinal disorders) | 37 | 44 | 0
Nausea (Gastrointestinal disorders) | 42 | 40 | 1
Vomiting (Gastrointestinal disorders) | 39 | 35 | 0
Asthenia (General disorders) | 31 | 27 | 0
Fatigue (General disorders) | 84 | 90 | 1
Oedema Peripheral (General disorders) | 61 | 55 | 2
Influenza (Infections and infestations) | 42 | 20 | 3
Nasopharyngitis (Infections and infestations) | 47 | 36 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 42 | 29 | 2
Urinary Tract Infection (Infections and infestations) | 39 | 20 | 3
Alanine Aminotransferase Increased (Investigations) | 100 | 77 | 5
Aspartate Aminotransferase Increased (Investigations) | 91 | 68 | 5
Blood Lactate Dehydrogenase Increased (Investigations) | 40 | 32 | 1
Weight Increased (Investigations) | 54 | 51 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 23 | 33 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 83 | 72 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 143 | 23 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 96 | 86 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 120 | 122 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 81 | 90 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 32 | 42 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 72 | 69 | 2
Headache (Nervous system disorders) | 46 | 31 | 2
Insomnia (Psychiatric disorders) | 32 | 30 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 18 | 2
Hot Flush (Vascular disorders) | 92 | 76 | 1
Hypertension (Vascular disorders) | 229 | 133 | 4

LIMITATIONS AND CAVEATS:
As per protocol the long-term extension (LTE) phase was planned but LTE phase is not included as part of this study hence no data was reported for LTE phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.